CLINICAL TRIAL: NCT04153357
Title: Comparison of Airtraq and C-mac in Pediatric Patients Under 1 Year Old
Brief Title: Comparison of Different Video Laryngoscopes in < 1 Year Old Undergoing Neurosurgical Operations: a Prospective Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Zehra Ipek ARSLAN, Associate Professor, Kocaeli University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: KOU KAEK 2016/315
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Intubation;Difficult
Keywords: airtraq; c-mac; videolaryngoscope; infant; intubatioon

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intubation time airtraq (Active Comparator): intubation time of Airtraq
  Interventions: Device: airtraq
- intubation time of c-mac (Active Comparator): intubation time of c-mac
  Interventions: Device: c-mac

INTERVENTIONS:
Device: airtraq — device entering the oral cavity till visualization of the endotracheal tube entering the vocal cords
  Other Names: videolaryngoscope
  Arms: intubation time airtraq
Device: c-mac — device entering the oral cavity till visualization of the endotracheal tube entering the vocal cords
  Other Names: videolaryngoscope
  Arms: intubation time of c-mac

SUMMARY:
İntubation of pediatric patients is a challenging problem. Video laryngoscopes increased the intubation success rate. We want to compare different video laryngoscopes in this field.

DETAILED DESCRIPTION:
Aim:İntubation of pediatric patients is a challenging problem. Video laryngoscopes increased the intubation success rate. We want to compare different video laryngoscopes in this field.

methods: We enroll total 50 patients < 1 year old undergoing neurosurgery. We compared the intubation times, success rates and minor complications of Airtraq and c-mac video laryngoscopes in these pediatric patients undergoing neurosurgery.

ELIGIBILITY:
Inclusion Criteria:

< 1 years old

* undergoing neurosurgery ASA 1-2

Exclusion Criteria:

* > 1 year old
* asa 3-4
* emergency

Ages: 1 Month to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
intubation time | 30 seconds
  device entering the oral cavity till visualization of the endotracheal tube entering the vocal cords

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University Medical Faculty, Kocaeli, Turkey (Türkiye)